CLINICAL TRIAL: NCT03728023
Title: A Phase I, Randomized, Double Blind, Placebo Controlled 2-Parts Study to Assess the Safety, Tolerability, Pharmacokinetics of AZD4205 Following Single and Multiple Ascending Dose in Healthy Adult Subjects, and to Assess the Effect of Food on the Pharmacokinetics of AZD4205
Brief Title: A Study of AZD4205 in Healthy Adult Subjects
Acronym: JACKPOT2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DZ2018J0001
Record Dates: First submitted 2018-10-28; First posted 2018-11-01 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2019-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD4205 (Experimental): Single ascending dose: 5mg, 20mg, 50mg, 100mg, 150mg Multiple ascending dose: low, medium and high dose once daily X 14 days
  Interventions: Drug: AZD4205
- Placebo (Placebo Comparator): placebo single dose in SAD and once daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4205 — SAD: 5mg, 20mg, 50mg, 100mg and 150mg MAD: low, medium and high dose once daily X14 days
  Arms: AZD4205
Drug: Placebo — Single dose in SAD and once daily for 14 days
  Arms: Placebo

SUMMARY:
This study is to assess the safety, tolerability, pharmacokinetics of AZD4205 following single and multiple ascending dose in healthy adult subjects, and to assess the effect of food on the pharmacokinetics of AZD4205.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to understand the nature of the trial and provide a signed and dated, written informed consent form prior to any study specific procedures, sampling and analyses.
2. Female and/or male aged ≥18 ~ ≤ 45 years, with BMI ≥18~≤ 28kg/m2.
3. Female subjects must have negative pregnancy tests at screening and check-in AND: have been surgically sterile OR post-menopausal OR, if of child-bearing potential, must be using an acceptable method of contraception.
4. Male subjects must be surgically sterile or using an acceptable method of contraception during the study and for 6 months after the last dose of AZD4205 or matching placebo to prevent pregnancy with a partner.

Exclusion Criteria:

1. Evidence or reported history of clinically significant hematological (absolute neutrophil count < 1.5 x 10^3/μL; platelet count < 100 x 10^3/μL; hemoglobin < 9 g/dL, INR > 1.5), renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease determined by the investigator.
2. Infections
3. Received a live vaccine within 3 months before first dose of IP.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
The number of subjects with adverse events | From screening up to 28 days after last dose (day29 for MAD, day 43 for food effect, day 42 for MAD)
  To evaluate the safety and tolerability of AZD4205 versus placebo in healthy subjects at different dose levels in terms of adverse events (AEs)
The number of subjects with abnormal laboratory parameters | From screening up to 28 days after last dose (day29 for MAD, day 43 for food effect, day 42 for MAD)
  To evaluate the safety and tolerability of AZD4205 versus placebo in healthy subjects at different dose levels in terms of abnormal laboratory parameters
The number of subjects with abnormal vital signs | From screening up to 28 days after last dose (day29 for MAD, day 43 for food effect, day 42 for MAD)
  To evaluate the safety and tolerability of AZD4205 versus placebo in healthy subjects at different dose levels in terms of abnormal vital signs
The number of subjects with abnormal electrocardiogram | From screening up to 28 days after last dose (day29 for MAD, day 43 for food effect, day 42 for MAD)
  To evaluate the safety and tolerability of AZD4205 versus placebo in healthy subjects at different dose levels in terms of abnormal electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Tracey, Principal Investigator — Frontage Clinical Services, Inc.
Locations (1):
- Frontage clinical service, Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen K, Guan X, Yang Z, Zhou Y, Liu Z, Deng X, Liu D, Hu P, Chen R. Pharmacokinetic characteristics of golidocitinib, a highly selective JAK1 inhibitor, in healthy adult participants. Front Immunol. 2023 Apr 3;14:1127935. doi: 10.3389/fimmu.2023.1127935. eCollection 2023. PMID 37077916